CLINICAL TRIAL: NCT01046188
Title: Development of an Interactive Web-based Teaching Tool for IVF Patients
Brief Title: Development of an Interactive Web-based Teaching Tool for in Vitro Fertilization (IVF) Patients
Acronym: WebIVF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Fertility Centre (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Dr Tannys Vause, Ottawa Fertility Centre
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: OFC01
Record Dates: First submitted 2010-01-07; First posted 2010-01-11 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Education
Keywords: Education; Internet; In vitro fertilization
MeSH Terms: interventions — Perceived Stress Scale

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Web-based Teaching Group (Experimental): Patients randomized to the intervention group will receive a unique login and password to a link on the Ottawa Fertility Centre website. This will allow them access to a secure site containing required teaching modules. They will then complete an interactive teaching tool that contains the same educational content as the traditional presentation. Patients will be able to access a module that is specific to their stimulation protocol. The teaching tool does not need to be completed all at one time. Once completed, the information can still be accessed as many times as required.
  Interventions: Other: Knowledge Questionnaire; Other: Perceived Stress Scale; Other: Satisfaction questionnaire; Other: Web-based IVF teaching
- Control group (Active Comparator): Participants randomized to the control arm of the study will participate in a traditional didactic teaching session. This session will be carried out by the nurse educator. This session will be attended by up to 10 other couples that may or may not be participating in the study. The nurse educator administering the session will not know which couples are participating in the study. Slides shown and information conveyed will be the same as that provided to the web-based group, however all three stimulation protocols will be presented to the participants regardless of their actual treatment protocol.
  Interventions: Other: Knowledge Questionnaire; Other: Perceived Stress Scale; Other: Satisfaction questionnaire; Other: Didactic lecture

INTERVENTIONS:
Other: Knowledge Questionnaire — Administered before and after teaching intervention
Other: Perceived Stress Scale — Administered before and after teaching intervention
Other: Satisfaction questionnaire — Administered after the intervention and at study completion
Other: Web-based IVF teaching — Web-based IVF teaching
  Arms: Web-based Teaching Group
Other: Didactic lecture — Didactic lecture
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate an interactive web-based teaching tool in IVF patients. Patients will be randomized to participate in web-based IVF teaching or a didactic lecture. A knowledge questionnaire will be completed both prior to and following the teaching intervention. Both groups will also complete stress and satisfaction surveys throughout the IVF treatment cycle. Groups will be compared at the completion of the study for demographics, level of knowledge, stress and satisfaction. The web-based group will be evaluated for web usage.

ELIGIBILITY:
Inclusion Criteria:

* Subject >18 years of age
* Able to provide informed consent
* First cycle of IVF
* English speaking and reading
* Internet access at home or work (that is easily accessible for personal use)

Exclusion Criteria:

* Failure to complete a baseline knowledge questionnaire prior to IVF consent signing
* Previous attendance at an IVF teaching session
* Previous IVF treatment (at the Ottawa Fertility Centre or any other IVF clinic)
* Undergoing Natural Cycle IVF (these patients do not generally participate in teaching sessions, as they undergo one-on-one teaching)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-01

PRIMARY OUTCOMES:
To assess knowledge in IVF patients after completing either a web-based teaching module or traditional teaching session | Assessed prior to consenting to IVF treatment and after teaching intervention (within 6-8 weeks)

SECONDARY OUTCOMES:
To assess stress levels in IVF patients after completing either a web-based teaching module or traditional teaching session | Assessed prior to consenting to IVF treatment and after teaching intervention (within 6-8 weeks)
To assess satisfaction in IVF patients after completing either a web-based teaching module or traditional teaching session | Assessed after the teaching intervention and at study completion (within 4-6 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Tannys DR Vause, MD, Principal Investigator — Ottawa Fertility Centre, University of Ottawa; Jason K Min, MD, Study Director — Ottawa Fertility Centre, University of Ottawa; Mark Evans, MBA, Study Director — Ottawa Fertiilty Centre
Locations (1):
- Ottawa Fertility Centre, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Haagen EC, Tuil W, Hendriks J, de Bruijn RP, Braat DD, Kremer JA. Current Internet use and preferences of IVF and ICSI patients. Hum Reprod. 2003 Oct;18(10):2073-8. doi: 10.1093/humrep/deg423. PMID 14507823
- [Background] Zebrack JR, Mitchell JL, Davids SL, Simpson DE. Web-based curriculum. A practical and effective strategy for teaching women's health. J Gen Intern Med. 2005 Jan;20(1):68-74. doi: 10.1111/j.1525-1497.2005.40062.x. PMID 15693931
- [Background] Kerfoot BP, Brotschi E. Online spaced education to teach urology to medical students: a multi-institutional randomized trial. Am J Surg. 2009 Jan;197(1):89-95. doi: 10.1016/j.amjsurg.2007.10.026. Epub 2008 Jul 9. PMID 18614145
- [Background] Ochoa JG, Wludyka P. Randomized comparison between traditional and traditional plus interactive Web-based methods for teaching seizure disorders. Teach Learn Med. 2008 Apr-Jun;20(2):114-7. doi: 10.1080/10401330801989513. PMID 18444196
- [Background] Nilsson M, Bolinder G, Held C, Johansson BL, Fors U, Ostergren J. Evaluation of a web-based ECG-interpretation programme for undergraduate medical students. BMC Med Educ. 2008 Apr 23;8:25. doi: 10.1186/1472-6920-8-25. PMID 18430256
- [Background] Spagnoletti CL, Sanders AM, McGee JB, Bost JE, McNeil MA. Teaching internal medicine residents to care for reproductive-age and pregnant women: an effective Web-based curriculum. Teach Learn Med. 2008 Apr-Jun;20(2):186-92. doi: 10.1080/10401330801991907. PMID 18444208
- [Background] Huang JY, Al-Fozan H, Tan SL, Tulandi T. Internet use by patients seeking infertility treatment. Int J Gynaecol Obstet. 2003 Oct;83(1):75-6. doi: 10.1016/s0020-7292(03)00253-4. No abstract available. PMID 14511879